CLINICAL TRIAL: NCT04817748
Title: Metabolomics Characterization of Biomarkers of Different Types of Myocardial Infarction in Different Time.
Acronym: MCBDTMIDT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, cardiology department of shanghai 10th people's hospital, Shanghai 10th People's Hospital
Other Study IDs: MCBDTMIDT
Record Dates: First submitted 2021-03-13; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Infarction
Keywords: myocardial infarction; metabolomics; biomarkers
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood extract plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Acute ST segment elevation myocardial infarction（STEMI）: the patients' coronary and venous blood were drawn for metabolomics study
- Acute non ST segment elevation myocardial infarction（NSTEMI）: the patients' coronary and venous blood were drawn for metabolomics study
- Acute myocardial infarction with no obstructive coronary atherosclerosis（MINOCA）: the patients' coronary and venous blood were drawn for metabolomics study
- Patients with normal coronary artery（NCA): the patients' coronary and venous blood were drawn for metabolomics study

SUMMARY:
To find new biomarkers through Metabonomics Study of different types of myocardial infarction in Different Time.

DETAILED DESCRIPTION:
In recent years, with the deepening understanding of the mechanism of myocardial infarction, in addition to the early understanding of plaque rupture, plaque erosion and other mechanisms, studies have found that inflammation, immunity, metabolism and other factors also play an increasingly important role in the occurrence and development of myocardial infarction. The LoDoCo2 study published at the 2020 ESC annual meeting and the COLCOT study previously published confirmed for the first time the therapeutic effect of anti-inflammatory drug colchicine in chronic coronary disease and acute myocardial infarction. At the same time, the fourth international definition of myocardial infarction also defines three different types of acute ST segment elevation myocardial infarction (STEMI), acute non ST segment elevation myocardial infarction (NSTEMI) and non infarct acute myocardial infarction (MINOCA). However, there are no clear research results on the mechanism, especially the mechanism of MINOCA. Therefore, the study of acute myocardial infarction in three groups is of great significance.

ELIGIBILITY:
Inclusion Criteria:

1.The patient clearly had acute myocardial infarction. 2.The patient's serum cardiac markers (mainly troponin) were elevated (at least above the upper limit of 99% reference value) and accompanied by one of the following clinical indicators：

1. Ischemic symptoms
2. New ischemic ECG changes, new ST-T changes or left bundle branch block（LBBB）.
3. Pathological Q wave formation in ECG
4. Imaging evidence showed new loss of myocardial activity or new regional wall motion abnormalities.
5. The thrombus was confirmed by coronary angiography. 3．The patient had chest pain symptoms, but coronary angiography showed normal coronary artery (such as intercostal neuralgia, cervical spondylosis, chest pain of unknown origin, etc.)

Exclusion Criteria:

1. Refusal to sign informed consent.
2. Surgical treatment was performed in the last three months.
3. Patients with a history of the following diseases or consider the diagnosis of the following diseases：Stress cardiomyopathy, myocarditis, pericarditis, pneumonia, pulmonary embolism, aortic dissection.
4. Severe heart failure, grade IV cardiac function.
5. Liver and kidney dysfunction.
6. blood-borne diseases, including HIV / AIDS, hepatitis B, hepatitis C, etc.
7. Patients with a history of malignancies, autoimmune diseases, severe infectious diseases and trauma.
8. Previous history of myocardial infarction and stroke.

Ages: 20 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Different types of myocardial infarction were identified according to the international definition of myocardial infarction and 2020 guidelines and consensus on myocardial infarction.
  2. Patients with normal coronary arteries were determined according to the results of coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
metabolites molecules | 6 months
  Detection of small molecular metabolites in blood by liquid chromatography mass spectrometry and gas chromatography mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhang, MD, Principal Investigator — Department of Cardiology, Shanghai Tenth People's Hospital
Locations (1):
- Yi Zhang, Shanghai, Shanghai Municipality, China